CLINICAL TRIAL: NCT01559571
Title: Study Registry for Severe Retinopathy and Treatment on Visual Outcomes of Premature Neonates
Brief Title: Registry for Severe ROP and Treatment on Visual Outcomes
Status: Completed | Type: Observational
Sponsor: Pediatrix (Other)
Responsible Party: Sponsor
Other Study IDs: PDX-01-011
Record Dates: First submitted 2012-02-28; First posted 2012-03-21 (Estimated); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Retinopathy of Prematurity
Keywords: Retinopathy of Prematurity
MeSH Terms: conditions — Retinopathy of Prematurity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine what factors influence the visual outcomes of infants with severe retinopathy of prematurity (ROP) and to monitor the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of informed consent and authorization
* Inborn and those admitted within 7 days of birth
* Infant with a diagnosis of stage 2 ROP or higher
* Site ability to plan close ophthalmological follow-up due to significant and persistent ROP
* Parents must agree to report outcomes following each ophthalmological visit and overall outcomes for up to five (5) years of age
* Ability to obtain follow-up data on outcomes if the child is transferred to another facility
* No known major congenital anomalies

Exclusion Criteria:

* ROP stage 1 or less
* Parents unwilling to participate in follow-up
* Major congenital anomalies

Max Age: 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Neonates who have a diagnosis of Retinopathy of Prematurity Stage 2 or higher
Sampling Method: Non-Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2012-05; Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Identification of visual acuity in subjects who were treated for ROP | Five year follow-up

SECONDARY OUTCOMES:
Recurrence of stage 3+ retinopathy of prematurity in one or both eyes in zone I or posterior zone II Recurrence of stage 3+ retinopathy of prematurity in one or both eyes in zone I or posterior zone II | Five year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Reese H Clark, MD, Principal Investigator — Pediatrix
Locations (2):
- United States (2):
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Summerlin Hospital Medical Center, Las Vegas, Nevada

REFERENCES:
- [Derived] Tolia VN, Ahmad KA, Jacob J, Kelleher AS, McLane N, Arnold RW, Clark RH; MEDNAX ROP Registry Investigators. Two-Year Outcomes of Infants with Stage 2 or Higher Retinopathy of Prematurity: Results from a Large Multicenter Registry. Am J Perinatol. 2020 Jan;37(2):196-203. doi: 10.1055/s-0039-1694983. Epub 2019 Sep 3. PMID 31480086